CLINICAL TRIAL: NCT05940701
Title: The Effectiveness of Biomimetic Materials in Preventing Enamel Demineralization During Fixed Appliance Orthodontic Treatment: a Randomized Clinical Trial
Brief Title: The Effectiveness of Biomimetic Materials in Preventing Enamel Demineralization During Fixed Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Samar Husam Assim, Orthodontics master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 763423
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Enamel Hypomineralization, Dental
MeSH Terms: conditions — Dental Enamel Hypomineralization | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive Curasept toothpaste with instructions and additionally at each visit a Curasept Biosmalto Mousse will be applied on the facial surface of the maxillary and mandibular anterior teeth using a tray.
  Interventions: Combination Product: Curasept Biosmalto Mousse and toothpaste
- control group (Placebo Comparator): The control group will receive a fluoridated toothpaste (Colgate toothpaste) and instructed to brush at least three times/day.
  Interventions: Other: Colgate toothpaste

INTERVENTIONS:
Combination Product: Curasept Biosmalto Mousse and toothpaste — at each visit a Curasept Biosmalto Mousse will be applied on the facial surface of the maxillary and mandibular anterior teeth using a tray.
  Arms: intervention group
Other: Colgate toothpaste — The control group will receive a fluoridated toothpaste (Colgate toothpaste)
  Arms: control group

SUMMARY:
This study will be done to evaluate the impact of Biosmalto Impact Action Mousse™ on the development and healing of WSLs in individuals receiving orthodontic treatment.

The control group received a fluoridated toothpaste (Colgate toothpaste). The intervention group received Curasept toothpaste and additionally at each visit a Curasept Biosmalto Mousse was applied on the facial surface of the maxillary and mandibular anterior teeth using a tray.

For each patient recruited, identical toothbrushes and oral care instructions were given. The patients received instructions to brush their teeth for at least two minutes using an up-down motion on their anterior teeth and a circular motion on their posterior teeth at least three times/day.

DETAILED DESCRIPTION:
This study is a multicenter randomized clinical trial with blinded parallel groups, simple randomization, an equal allocation ratio (1:1), and no stratification.The patients will be initially assessed for eligibility to be included in the study by the investigator.The study was verbally explained to those who fulfilled the inclusion criteria in order to get their first consent for participation. After that, they received the patient information sheet (Appendix), which explained the purpose of the research. The patients were instructed to thoroughly read the informational material at home and tell the researcher of their intention to participate at the next visit. Participants had to either sign the consent form (which was attached to the patient information sheet) or get their parents' permission (if the participant was under the age of 18 years). The investigator provided the patients with further information or reassurance about the trial if needed.

All the participants received a standardized treatment protocol. The patients were treated with straight wire appliance using metal brackets (3BOrtho, China). Initially, teeth polishing was performed with pumice and rubber cup for 10 seconds using a low-speed handpiece, followed by water rinsing and air drying (oil-free air spray for 30 seconds). Bonding technique was performed using 37% phosphoric acid for 30 seconds (Heinig and Hartmann, 2008b), then washed with water for 15-20 seconds, and dried for 10 seconds. A thin coat of primer was applied to the etched surfaces by an applicator and cured for 15 seconds by the LED light-curing unit. The brackets were bonded using similar adhesive (3B Ortho, white glue, China) and checked so that no obvious extra adhesive is remained on the tooth surface around the brackets. The control group received a fluoridated toothpaste (Colgate toothpaste). The intervention group received Curasept toothpaste and additionally at each visit a Curasept Biosmalto Mousse was applied on the facial surface of the maxillary and mandibular anterior teeth using a tray.

For each patient recruited, identical toothbrushes and oral care instructions were given. The patients received instructions to brush their teeth for at least two minutes using an up-down motion on their anterior teeth and a circular motion on their posterior teeth at least three times/day. Additionally, the patients were instructed not to use any additional antimicrobial-containing products (mouthwash, toothpaste, gel).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate.
* No underlying medical conditions requiring medications that may cause dryness of the mouth.
* Fully erupted permanent maxillary and mandibular canines and incisors that have not been restored.

Exclusion Criteria:

* Receiving professional fluoridation within the last three months.
* Untreated cavitated lesions or significant restorations on the facial surfaces of study teeth.
* Labial restoration of any of the study teeth.
* Missing any of the study teeth.
* Severely rotated any of the study teeth (limiting the appearance of buccal surfaces).
* Patients with enamel hypoplasia, dental fluorosis or tetracycline pigmentation.
* Dental anomalies related to morphology, anatomy, or development.
* Pregnancy and xerostomia.
* Heavy smokers.
* Craniofacial syndromes such as clefts

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
WSLs evaluation | 6 month
  To evaluate the number of WSLs on the labial surfaces of maxillary and mandibular anterior teeth using enamel white spot lesion index (WSLI), ICDAS (International caries detection and assessment system) and DIAGNOdent pen scores at each visit and after six months during orthodontic treatment.
  Gorelick Index :
  0: no WSLs
  1. Slight WSLs
  2. extended or excessive WSLs
  3. WSLs with cavitation
  DIAGNOdent pen reading:
  0 - 10 Healthy Tooth Structure 11-20 Outer Half Enamel Caries 21-30 Inner Half Enamel Caries 30+ Dentin Caries

SECONDARY OUTCOMES:
amount of plaque and gingival bleeding | 6 month
  To evaluate the amount of plaque and gingival bleeding by using visible plaque index (VPI) gingival bleeding index (GBI) at each visit (4-6 weeks) Visible plaque index (VPI) 0: non-visible plaque 1: visible plaque Gingival bleeding index (GBI) 0: no gingival bleeding
  1: gingival bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Husam Assim Alkhdhairi, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson A, Skold-Larsson K, Hallgren A, Petersson LG, Twetman S. Effect of a dental cream containing amorphous cream phosphate complexes on white spot lesion regression assessed by laser fluorescence. Oral Health Prev Dent. 2007;5(3):229-33. PMID 17977295
- [Background] Ardu S, Castioni NV, Benbachir N, Krejci I. Minimally invasive treatment of white spot enamel lesions. Quintessence Int. 2007 Sep;38(8):633-6. PMID 17823680
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] Cosma LL, Suhani RD, Mesaros A, Badea ME. Current treatment modalities of orthodontically induced white spot lesions and their outcome - a literature review. Med Pharm Rep. 2019 Jan;92(1):25-30. doi: 10.15386/cjmed-1090. Epub 2019 Jan 15. PMID 30957083
- [Background] Du J, Yuan Y, Si T, Lian J, Zhao H. Customized optimization of metabolic pathways by combinatorial transcriptional engineering. Nucleic Acids Res. 2012 Oct;40(18):e142. doi: 10.1093/nar/gks549. Epub 2012 Jun 19. PMID 22718979
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Gizani S, Kloukos D, Papadimitriou A, Roumani T, Twetman S. Is Bleaching Effective in Managing Post-orthodontic White-spot Lesions? A Systematic Review. Oral Health Prev Dent. 2020 Feb 14;18(1):2-10. doi: 10.3290/j.ohpd.a44113. PMID 32051965
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Iafisco M, Degli Esposti L, Ramirez-Rodriguez GB, Carella F, Gomez-Morales J, Ionescu AC, Brambilla E, Tampieri A, Delgado-Lopez JM. Fluoride-doped amorphous calcium phosphate nanoparticles as a promising biomimetic material for dental remineralization. Sci Rep. 2018 Nov 19;8(1):17016. doi: 10.1038/s41598-018-35258-x. PMID 30451901
- [Background] Sonesson M, Bergstrand F, Gizani S, Twetman S. Management of post-orthodontic white spot lesions: an updated systematic review. Eur J Orthod. 2017 Apr 1;39(2):116-121. doi: 10.1093/ejo/cjw023. PMID 27030284
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Derived] Assim SH, Yassir YA. Effect of biomimetic tooth mousse and toothpaste on the incidence of white spot lesions during fixed appliance orthodontic treatment: A randomized clinical trial. J Taibah Univ Med Sci. 2025 Jun 25;20(3):405-416. doi: 10.1016/j.jtumed.2025.06.004. eCollection 2025 Jun. PMID 40657473